CLINICAL TRIAL: NCT01406600
Title: Optimal rhCG(Ovidrel®) Dose for Final Oocyte Maturation Triggering in Poor Responder During IVF and ICSI Cycles
Brief Title: Optimal rhCG(Ovidrel®) Dose in Poor Responder During IVF and ICSI Cycles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Seok Hyun Kim, Seok Hyun Kim, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hCG dose_oocyte maturity
Record Dates: First submitted 2011-07-23; First posted 2011-08-01 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: in Vitro Fertilization; Poor Responder
Keywords: recombinant hCG; poor responder; oocyte maturity
MeSH Terms: interventions — Ovidrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- rhCG 250mcg (Active Comparator): For final oocyte maturation triggering in ART, rhCG 250mcg will be administrated.
  Interventions: Drug: recombinant hCG (Ovidrel®)
- rhCG 500mcg (Experimental): For final oocyte maturation triggering in ART, rhCG 500mcg will be administrated.
  Interventions: Drug: recombinant hCG (Ovidrel®)

INTERVENTIONS:
Drug: recombinant hCG (Ovidrel®) — Recombinant hCG (Ovidrel®)will be administrated for final oocyte maturation triggering in poor responders with different two doses (250mcg vs. 500mcg). Usually rhCG is administrated after 24~48 hours from optimal ovarian stimulation status.

SUMMARY:
Choriogonadotropin alfa (Ovidrel®) is a recombinant hCG (rhCG) preparation derived from genetically engineered Chinese hamster ovary cells, which is widely used for final oocyte maturation triggering in assisted reproductive technology (ART).Recombinant hCG has been investigated about its safety and efficacy comparing with urinary hCG, but still the optimal dose of rhCG is questionable. From former studies, there only have been proven that high dose of hCG can make ovarian hyperstimulation syndrome (OHSS) in usual condition. On the other hand, we hypothesize that high dose of hCG may improve oocyte maturity in poor responders who cannot easily provoke OHSS. Hence, this study will assess the comparative efficacy and safety of 250mcg and 500mcg of rhCG in ART treatment cycle.

DETAILED DESCRIPTION:
Randomized prospective clinical study that compare the two doses of rhCG (250mcg vs. 500mcg).

ELIGIBILITY:
Inclusion Criteria:

* poor response in prior IVF cycle (≤ 4 oocyte retrieved)
* women's age ≥ 40 years
* FSH ≥ 10mIU/mL or AMH ≤ 1.1ng/mL
* Antral follicle count <6

Exclusion Criteria:

* patient without informed consent

Ages: 21 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-11 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
oocyte maturity | Up to the ovum pick up day. At the point of ovum pick-up, we can count how many mature or immature oocytes were retrived. Therefore, in one hour after ovum pick-up, outcome measurement will be possible.
  After administration of different doses of rhCG, oocyte maturity will be assessed on ovum pick up day. Oocytes will be classified into GV, MI, and MII.

SECONDARY OUTCOMES:
clinical pregnancy rate | After confirming fetal heart beat via transvaginal ultrasound. Usually 2 to 4 weeks after ovum pick-up day.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea